CLINICAL TRIAL: NCT05585658
Title: A Randomized, Double-blinded, Active Controlled, Single Dosing, Crossover Clinical Trial to Investigate the Pharmacokinetics, Pharmacodynamics and Safety of GBPD002 and Eprex® After Subcutaneous Administration in Healthy Adult Volunteers.
Brief Title: A Randomized, Double-blinded, Active Controlled Crossover Clinical Trial to Investigate PK, PD and Safety of GBPD002
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Globe Biotech Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DGDA/CTP-1/06/2016/9916
Record Dates: First submitted 2022-09-25; First posted 2022-10-19 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Natural Blood and Blood Product Toxicity
Keywords: human recombinant erythropoietin
MeSH Terms: interventions — Epoetin Alfa

STUDY DESIGN:
Intervention Model Description: Healthy volunteers participating in two cohorts. In each cohort 21 volunteers are participating in the clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the objectives of the study, the identity of test and control treatments will not be known to investigators, research staff, or subjects. The following study procedures will be in place to ensure double-blind administration of study treatments. Blinded (investigators) and unblinded (study nurses responsible for administration of study medication) study personnel had to be involved in order to preserve blinding of the investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erythropoietin alpha Eprex® (Active Comparator): Group/cohort/Arm 1 (participating 21 volunteers): Eprex® injection 4,000 IU will be administered subcutaneously on Day 1; and wash out for 4 weeks. GBPD002 injection 4,000 IU/1 mL will be administered subcutaneously on Day 29.
  Interventions: Biological: Erythropoietin alpha
- Erythropoietin alpha, GBPD002 (Experimental): Group/cohort/Arm 2 (participating 21 volunteers):GBPD002 PFS (Pre-Filled Syringe) 4,000 IU/ 1 mL (Erythropoietin alfa 4,000 IU) will be administered subcutaneously on Day 1.And wash out for 4 weeks (28 days from the 1st injection day). Eprex® inj. (Injection) 4,000 IU (Erythropoietin alfa 4,000 IU) will be administered subcutaneously on Day 29.
  Total 42 volunteers participated in the clinical trial.
  Interventions: Biological: Erythropoietin alpha

INTERVENTIONS:
Biological: Erythropoietin alpha — To analyze bio-similarity of GBPD002 with Eprex®, the Globe Biotech Ltd performed quite a few experiments to determine total analytical study of GBPD002. They performed peptide mapping to determine amino acid composition of GBPD002 and found similar result with erythropoietin alpha. The molecular weight was determined through SDS-PAGE analysis of GBPD002 and was compared with Eprex. The western blot analysis was performed to determine immune chemical characterization. Characterization of different isoforms was conducted through 2D gel electrophoresis.

SUMMARY:
Erythropoietin (EPO) biosimilarity for GBPD002 (test candidate) and Eprex® (comparator) has been evaluated by comparing the pharmacokinetic (PK) and pharmacodynamic (PD) properties following subcutaneous injection in human subjects. This was a randomized, double-blind, two-sequence, crossover study. Subjects were randomly assigned and received a dose (4,000 IU) of either the test or comparator EPO. The subjects received the alternative formulation after the wash out period (4 weeks) of the first administration. The primary PK parameters, viz., maximum observed concentration (Cmax) and area under the curve extrapolated to infinity (AUC00-inf), were calculated with the serum EPO concentrations from blood samples and were found comparable for both formulations. The geometric mean ratios (@90% CI) of the Cmax and AUCinf were 1.16 and 0.89, respectively, which were within the regulatory range of 0.80-1.25. The reticulocyte, hematocrit, hemoglobin and red blood cell counts were measured as PD markers. The time-matched serum EPO concentrations and PD markers denoted a counterclockwise hysteresis, and thereby suggesting a time delay between the observed concentration and the response. ANOVA derived P-values (all were greater than 0.05) for the effectors clearly revealed the similarity between effects on PD markers for both formulations. Both formulations were found tolerated well, and anti-drug antibodies were not observed. Thus, the two formulations are projected to be used interchangeably in clinical settings.

DETAILED DESCRIPTION:
Erythropoietin (EPO) is a glycoprotein hormone that plays a key role in the formation of red blood cells (RBCs). EPO is primarily synthesized in the peritubular cells of the kidney and released into the systemic circulation in adult individuals. Circulating EPO binds to the EPO receptor on bone marrow erythroid progenitors, triggering multiple signaling pathways that support differentiation into mature RBCs. A reduction in EPO production is the primary cause of anemia in people with chronic renal failure [4]. Human recombinant epoetin (rHuEPO) or erythropoiesis stimulating agents (ESA) have been demonstrated to stimulate erythropoiesis in anemic patients with chronic renal failure, including those who need and don't need dialysis. ESAs are used to treat chemotherapy-induced anemia in cancer patients and to reduce the requirement for allogenic blood transfusions in patients with mild anemia who are undergoing surgery. Furthermore, human recombinant epoetin is recommended for patients who are at high risk for perioperative transfusions due to considerable blood loss.

Recombinant rHuEPO was manufactured using recombinant DNA techniques. Alpha epoetins are the most commonly used type of rHuEPO among the other forms. Eprex®, the pioneer product of alpha epoetins, is a regular medicine with proven efficacy and tolerability. Globe Biotech Limited, a Bangladeshi biopharmaceutical company has developed GBPD002, a biosimilar of Eprex® which is synthesized in genetically engineered Chinese hamster ovary (CHO) cells. Upstream and downstream process development and validation was done for large scale production. Step by step identical analytical results confirmed the biosimilarity of GBP002 with Eprex®. Single and repeat dose toxicity was performed in Wister rat to analyze the toxicity of GBPD002 with Eprex®.

The aim of this study is to analyze the bioequivalence of GBPD002 and Eprex®. The purpose of this study is to compare the pharmacokinetic (PK), pharmacodynamics (PD) and safety of human recombinant erythropoietin, GBPD002, developed by Globe Biotech Limited and the reference product Eprex® manufactured by Janssen Cilag Ltd., UK in healthy volunteers. An independent ethics committee gave ethical clearance for this study and the protocol for this study was approved by the Directorate General of Drug Administration (DGDA) of Bangladesh.

A randomized, double-blind, single-dose, and two-sequence crossover trial was conducted in 42 healthy volunteers in 2 groups/cohorts/arms. The Clinical Research Organization (CRO Ltd.) conducted this investigation at Farabi General Hospital, Dhanmondi R/A, Dhaka 1209, in compliance with the principles of the Declaration of Helsinki and the International Conference on Harmonization's Guideline for Good Clinical Practice. Bangladesh's Directorate General of Drug Administration (DGDA) approved the study methodology and informed consent form. Volunteers were given thorough information about the study and they have signed an informed consent form to affirm their willingness to participate.

The study was open to healthy male participants aged 19-45 years old who weighed 55.0-90.0 kg and had a body mass index of 18.0-27.0 kg/m2. Subjects were eliminated if they had at least one of the following clinical laboratory test results: Hemoglobin level <12 g/dL or >17 g/dL, vitamin B12 level <200 pg/mL, ferritin level <21.8 ng/mL, transferrin level <190 mg/dL and any anomalous range for the reticulocyte (RET) count, erythrocytes, platelets or serum potassium levels. The number of subjects was determined based on the results of a previous clinical study on a single subcutaneous injection of epoetin alfa in healthy subjects. The total number of subjects was 42, assuming a 20% dropout rate. COVID-19, HIV, HBsAg, and HCV (Hepatitis C Virus) positive individuals were excluded from the study.The recruited volunteers were randomly assigned to one of the two sequences and received a single subcutaneous injection of 4,000 IU of either the comparator drug (Eprex®) or the test drug (GBPD002) in the abdomen from a prefilled syringe (PFS), based on the allocated sequences with a 28-day washout period: sequence A, administered the comparator drug in period 1 followed by the test drug in period 2; sequence B, given the test drug in period 1 followed by the comparator drug in period 2.Blood samples were taken for the PK evaluation at predose and at 1, 3, 6, 8, 10, 14, 24, 48, 72, 96, 120 and 144 h postdose. For the PD evaluation, the reticulocyte count (RET; %), hematocrit (HCT; %), haemoglobin (HB) (g/L) and red blood cell (RBC) count (106/mm3) were calculated at predose and at 72, 144, 216, and 312 h postdose.

ELIGIBILITY:
Inclusion Criteria: The inclusion criteria of subjects for the study are following Healthy adults

* age:18 - 45 years;
* BMI:18.0 - 27.0 kg/m2;
* body weight: 55 - 90 kg;
* able to swallow tablets,
* clinically and mentally fit subjects having no comorbid disease condition such as ISD, heart failure, CKD, Alzheimer's diseases, liver cirrhosis.

Exclusion Criteria: Those whose results meet more than one of the following in the screening including re-test;

* Hemoglobin level below 12 g/dL or over 17g/dL,
* Vitamin B12 level below 200 pg/mL,
* Ferritin level below 21.8 ng/mL,
* Transferrin level below 190 mg/dL,
* Reticulocyte, erythrocytes,
* insulin dependent diabetes,
* Thyroid disease, platelets or serum potassium level over/below normal range.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The inclusion criteria of subjects for the study are following Age: 18 - 45 years; Body Mass Index (BMI): 18.0 - 27.0 kg/m2
Enrollment: 42 (Actual)
Dates: Start 2021-10-16 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Primary endpoint to measure safety, efficacy and acceptability of Erythropoietin medicine | 34 days
  EDTA-containing tube needs to be arranged for whole blood collection; for each test ~350 µL sample may require.Area under Curve last (AUC0-last) of Erythropoietin: Area Under Curve last (AUC0-last) of Erythropoietin [Time Frame: Once 1 hour before administration (day 1/day 29); 1, 3, 6, 8, 10, 14, 24, 48, 72, 96, 120, 144 (day 6/day 34) hrs after administration for each period]

SECONDARY OUTCOMES:
Secondary endpoints to measure safety, efficacy and acceptability of Erythropoietin medicine | 34 days
  EDTA-containing tubes need to be arranged for whole blood collection; for each test ~350 µL sample may require.Time of maximum concentration (Tmax) of Erythropoietin: Time of maximum concentration (Tmax) of Erythropoietin [Time Frame: Once 1 hour before administration (day 1/day 29); 1, 3, 6, 8, 10, 14, 24, 48, 72, 96, 120, 144 (day 6/day 34) hrs after administration for each period]

CONTACTS AND LOCATIONS:
Overall Officials: Mamun Al Mahtab, PhD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (2):
- Bangladesh (2):
  - Globe Biotech Limited, Dhaka
  - Farabi General Hospital, Dhaka

IPD SHARING:
Plan to Share IPD: No
We have NDA with volunteers to keep personal information's not to be published.